CLINICAL TRIAL: NCT07205601
Title: Phase 2a Assessment of Safety, Tolerability, and Efficacy of Repeated Dosing of Intracerebroventricular Injections of Ex Vivo Expanded, Autologous Adipose-Derived Stem Cells (RB-ADSCs) in Participants With Mild to Moderate Alzheimer's Disease
Brief Title: Study of Intracerebroventricular Injections of Autologous Adipose-Derived Stem Cells (RB-ADSCs) in Participants With Mild-Moderate Alzheimer's Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneration Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RB-ADSC-03
Record Dates: First submitted 2025-09-17; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease
Keywords: AD; Autologous; Stem cells; Cell therapy; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RB-ADSC low dose (Experimental): Participants will receive repeated doses of 2.5x10^6 RB-ADSC infused in the previously implanted Ommaya reservoir
  Interventions: Biological: RB-ADSC
- RB-ADSC high dose (Experimental): Participants will receive repeated doses of 5x10^6 RB-ADSC infused in the previously implanted Ommaya reservoir
  Interventions: Biological: RB-ADSC
- Placebo control (Placebo Comparator): Participants will receive placebo comparator in the previously implanted Ommaya reservoir
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: RB-ADSC — RB-ADSC is an investigational an ex-vivo expanded autologous adipose-derived stem cell product
  Arms: RB-ADSC high dose; RB-ADSC low dose
Other: Placebo — 0.9% NaCl USP
  Arms: Placebo control

SUMMARY:
The goal of this Phase 2 clinical trial is to learn if repeated dosing of RB-ADSC (an investigational autologous cell product obtained from participant's own adipose tissue) enhances the positive preliminary results seen in Phase 1 for the of treatment for mild to moderate Alzheimer's Disease in adults. The clinical trial will also continue to evaluate the safety of repeated dosing of RB-ADSC. This study will primarily evaluate the effects of repeated dosing of RB-ADSC on cognitive performance compared to placebo control. Participants will receive RB-ADSC every 2 months for a total of 6 doses. Participants randomized into the placebo control group will have the option to cross over to receive treatment after completion of the primary phase of the study.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, dose range finding for safety and efficacy, Phase 2a U.S. multicenter study of repeated administration of RB-ADSC in participants with mild to moderate Alzheimer's Disease AD. RB ADSC consists of stem cells obtained from the participant's own adipose tissue by lipoaspirate that have been cultured and expanded outside the body, enriched for Wnt-activated cells, and prepared for administration into the same participant. An Ommaya reservoir, which is an intraventricular catheter system, will be implanted under the scalp for intraventricular administration of RB-ADSC.

Approximately 115 adult participants are expected to be enrolled in this Phase 2a study. Participants will be randomized at a 4:1 ratio of RB-ADSC treatment to placebo. Participants randomized into the RB-ADSC treatment arm will be subsequently randomized with a 1:1 ratio to a treatment dose level: low-dose RB-ADSC (2.5 x 10^6 cells), and high-dose RB-ADSC (5.0 x 10^6 cells), for an overall randomization scheme of 2:2:1.

RB-ADSC will be delivered intracerebroventricularly every 2 months via the previously implanted Ommaya reservoir for a treatment duration of 10 months (inclusive of 10th month; up to 6 injections in total). Participants will be followed for 6 months after the last administration. The primary and secondary objectives will evaluate the efficacy based on cognitive, functional and CSF biomarker (Phospho-Tau, Total Tau, AB-42) assessments. Additionally, safety evaluations, volumetric MRI (Neuro Quant®) assessment, and diagnostic imaging comparison (Amyloid PET) will be performed.

After completing the Month 12 evaluation, participants in the placebo arm will be allowed to cross over to receive RB-ADSC. Participants in the cross-over will be randomized to a treatment dose level (low dose or high dose) at a 1:1 ratio. Cross-over participants will receive RB-ADSC doses every 2 months for a treatment duration of 10 months.

ELIGIBILITY:
Inclusion Criteria:

* ≥45 and ≤85 years of age
* Mild to moderate AD diagnosis
* FAST stage 4 or 5
* MMSE 10-23
* Amyloid PET scan centiloid score >30
* ADmark® CSF analysis of ATI (<1.0) and P-Tau (>60)
* No tumors or other disease responsible for dementia
* Participant otherwise in good general health
* Written informed consent from participant or legal representative
* Participant must have caregiver who separately meets specified inclusion/exclusion criteria for caregivers
* Participant must be able to donate adequate amount of lipoaspirate to establish the final product

Exclusion Criteria:

* Taking prohibited medications
* Prior cell therapy implantation
* Existing ventriculoperitoneal shunts
* Neurological disorders except AD
* Psychiatric disorders such as schizophrenia, bipolar/unipolar depression, delirium
* Drug or alcohol abuse in past 2 years
* History of cancer within the past 5 years
* No caregiver available to meet the inclusion criteria for caregivers
* Involvement in other investigational product clinical trial within the past 3 months for monoclonal antibodies, or 6 months for other investigational products

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline on the Integrated Alzheimer's Disease Rating Scale (iADRS) Composite Score | Baseline, Month 6 and Month 12
  iADRS will be used to assess whether RB-ADSC slows down the clinical decline associated with AD compared with placebo. iADRS evaluates cognition and daily function performance by combining items from the ADAS-Cog13 and the Alzheimer's disease cooperative study-instrumental activities of daily living scale (ADCS-iADL). The scale ranges from 0 to 144, where lower scores indicate worse performance and higher score indicates better performance.

SECONDARY OUTCOMES:
Change from Baseline in CSF Biomarkers | Baseline, Month 6 and Month 12
  CSF Biomarkers will be measured with the ADmark® phospho-tau/total-tau/ Abeta-42 assay to determine the levels of Phosphorylated-Tau protein, Total-Tau protein, and Ab42 in the cerebrospinal fluid (CSF). The amyloid-tau index (ATI) will also be determined.
Change from Baseline in MMSE | Baseline, Month 6 and Month 12
  Cognitive function will be evaluated with the Mini Mental State Examination (MMSE). The range for the total MMSE score is 0 to 30, with lower scores indicating greater level of impairment.
Change from Baseline in ADAS-cog13 | Baseline, Month 6 and Month 12
  Cognitive function will be assessed using the AD Assessment Scale - Cognitive (ADAS-cog13). The ADAS-Cog13 scale ranges from 0 to 85, with higher scores indicating greater disease severity.
Change from Baseline in FAST | Baseline, Month 6 and Month 12
  Functional abilities will be assessed using the Functional Assessment Staging Tool (FAST). The tool consists of seven stages, with higher scores indicating more severe impairment.
Change from Baseline in ADCS-iADL | Baseline, Month 6 and Month 12
  Functional ability will be assessed using the AD Cooperative Study-Activities of Daily Living Scale (ADCS-ADL). The iADL score ranges from 0 to 59, with lower scores indicating greater impairment.
Change from Baseline in CDR-SB | Baseline, Month 6 and Month 12
  Cognitive changes will be assessed with the Clinical Dementia Rating - Sum of Boxes (CDR-SB). Scores range from 0 to 18 with higher scores indicative of more impairment.
Change from Baseline in Amyloid Positron Emission Tomography (Amyloid-PET) | Baseline, Month 6 and Month 12
  Amyloid-PET will be used to quantitatively assess amyloid plaque deposition in the brain
Change from Baseline in Volumetric MRI with Contrast | Baseline, Month 6 and Month 12
  Volumetric MRI with contrast of the brain will be used to detect and monitor brain abnormalities.
Change from Baseline in NeuroQuant MRI | Baseline, Month 6 and Month 12
  NeuroQuant MRI will be used to measure volumes of brain structures.
Safety of Repeated Dosing RB-ADSC | Up to Month 16
  Safety will be determined by the number of treatment-related adverse events (AE) and serious adverse events (SAE) graded according to CTCAE v5.0 up to Month 16 compared to placebo control

IPD SHARING:
Plan to Share IPD: Undecided